CLINICAL TRIAL: NCT05937737
Title: The Effect of the Phytochemical Content and Total Antioxidant Capacity of the Diet on Serum FGF21 Levels in Type 2 Diabetes
Brief Title: Serum FGF21 Levels and Dietary Total Antioxidant Capacity in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GO 20/228
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
Keywords: FGF-21; type 2 diabetes; antioxidant capacity; phytochemical index
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 Diabetes (Experimental): Individuals with type 2 diabetes were followed for 12 weeks with an appropriate diet specific to their type 2 diabetes condition, and necessary measurements were taken at the beginning, 4th week, and 12th week.
  Interventions: Behavioral: Type 2 Diabetes Diet Modification
- Healthy Controls (No Intervention): No dietary intervention was made for the control group, and necessary measurements were taken at the beginning and 12th week.

INTERVENTIONS:
Behavioral: Type 2 Diabetes Diet Modification — A 12-week dietary intervention model was prescribed to the patients in accordance with their needs.
  Arms: Type 2 Diabetes

SUMMARY:
This study aimed to evaluate the phytochemicals and total antioxidant capacity in the diets of individuals with type 2 diabetes and assess their relationship with glycemic parameters, as well as certain biochemical parameters and Fibroblast growth factor 21 (FGF21), which is an inflammatory marker. The study was conducted on a total of 80 individuals, including 40 patients with overweight or obesity (Body Mass Index (BMI) > 25 kg/m²) with type 2 diabetes aged between 18 and 64, and 40 healthy controls (BMI between 18.5-35 kg/m²). The individuals were followed for 12 weeks with an appropriate diet. Biochemical parameters, anthropometric measurements, and dietary intake records were monitored at specific intervals throughout the study. The phytochemical index and total antioxidant capacity of the individuals' diets were measured, and FGF21 was examined in the serum.

DETAILED DESCRIPTION:
Individuals were divided into two groups: type 2 diabetes and control. Individuals with type 2 diabetes were followed for 12 weeks with an appropriate diet specific to their condition, and necessary measurements were taken at the beginning, 4th week, and 12th week. No dietary intervention was made for the control group, and necessary measurements were taken at the beginning and 12th week. At the control points, biochemical parameters, serum samples, anthropometric measurements (body composition, weight, height, waist circumference, hip circumference), 24-hour dietary intake record, and 24-hour physical activity record were evaluated. In the experimental group, dietary intake was recorded at the beginning (week 0), 4th week, and 12th week. The dietary intake of the control group was examined at week 0 and week 12.

The "Phytochemical Index" method was used to calculate the total phytochemical intake from the diet. The total antioxidant capacity of the diet was calculated using data obtained from dietary intake records based on Ferric Reducing Ability of Plasma (FRAP), Oxygen Radical Absorbance Capacity (ORAC), Trolox Equivalent Antioxidant Capacity (TEAC), and Total Reactive Antioxidant Potential (TRAP) methods. Additionally, physical activity was determined using a recording method. Body compositions at all three control points will be determined using the bioelectrical impedance method, and waist and hip circumference measurements were taken using a non-stretchable tape measure. Routine biochemical parameters for the type 2 diabetic group (fasting blood glucose, serum lipids, HbA1c) were obtained from the records. Serum samples collected after a 10-12 hour fasting period at the beginning and 12th week were analyzed for Fibroblast growth factor 21 (FGF21) using suitable kits.

ELIGIBILITY:
Inclusion Criteria:

* For intervention group: type 2 diabetes diagnosis
* For control group: healthy individuals
* Aged between 19 and 64
* With a body mass index over 25 kg/m²

Exclusion Criteria:

* Pregnancy
* Type 1 diabetes
* Cancer
* Chronic kidney disease
* Chronic liver disease
* Other chronic inflammatory diseases
* Individuals with HbA1c levels above 9%
* Individuals using short or medium-acting or mixed (medium+short) insulin
* Individuals with any condition that hinders physical activity
* Individuals following any weight loss diet

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Fibroblast growth factor 21 (FGF21) | 12 weeks
  FGF21 levels in serum
Body weight | 12 weeks
  Body weight measurements
Body fat percentage | 12 weeks
  Body fat percentage measured with bioelectrical impedance analysis
Phytochemical index | 12 week
  Dietary phytochemical index
Ferric Reducing Ability of Plasma (FRAP) | 12 weeks
  Dietary antioxidant capacity measured with FRAP method
Oxygen Radical Absorbance Capacity (ORAC) | 12 weeks
  Dietary antioxidant capacity measured with ORAC method
Trolox Equivalent Antioxidant Capacity (TEAC) | 12 weeks
  Dietary antioxidant capacity measured with TEAC method
Total Reactive Antioxidant Potential (TRAP) | 12 weeks
  Dietary antioxidant capacity measured with TRAP method

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Internal Medicine Department, Ankara
  - Hacettepe University Nutrition and Dietetics Department, Ankara

IPD SHARING:
Plan to Share IPD: No